CLINICAL TRIAL: NCT00002137
Title: A Phase I Trial of Tecogalan Sodium ( DS-4152 ) Administered as an Infusion Weekly x 4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 088B; 4152A-PRT002
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Neoplasms; Sarcoma, Kaposi; Acquired Immunodeficiency Syndrome; Antineoplastic Agents; tecogalan
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Neoplasms; Acquired Immunodeficiency Syndrome | interventions — tecogalan

INTERVENTIONS:
Drug: Tecogalan sodium

SUMMARY:
To evaluate the safety of different doses and dosing regimens of tecogalan sodium (DS-4152) and to establish the MTD at each of the different dosing schedules.

DETAILED DESCRIPTION:
Patients receive intravenous DS-4152 by infusion weekly for 4 weeks, followed by 2 weeks of rest; courses may repeat. Patients undergo weekly follow-up. A punch biopsy will be obtained from patients with Kaposi's sarcoma.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Kaposi's sarcoma plus HIV infection OR metastatic solid tumor.
* Life expectancy of at least 12 weeks.
* NO symptomatic AIDS-defining opportunistic infection within the past 4 weeks.
* Recovered from toxicity of any prior anticancer therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Leukemia or lymphoma.
* Current gastrointestinal bleeding by stool guaiac.
* Extensive bone metastases or significant radiographic osteoporosis in patients with solid tumors.
* Active heart disease such as uncontrolled angina, uncompensated congestive heart failure, or dysrhythmias requiring antiarrhythmics.
* Acute intercurrent infection other than genital herpes.
* Symptomatic or known central nervous system involvement (including brain metastases) unless stable and off therapy.

Concurrent Medication:

Excluded:

* Other anticancer therapy.
* Other investigational agents.

Patients with the following prior conditions are excluded:

* History of acute or chronic gastrointestinal bleeding or inflammatory bowel disease.
* History of myocardial infarction within past 6 months.

Prior Medication:

Excluded:

* Anticancer therapy within the past 3 weeks (6 weeks for nitrosourea or mitomycin C).
* Investigational agents within the past 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Kenneth Norris Jr Cancer Ctr / USC, Los Angeles, California, United States

REFERENCES:
- [Background] Tulpule A, Snyder JC, Espina BM, Higashi L, Satomi M, Lombardy EE. A phase I study of tecogalan, a novel angiogenesis inhibitor in the treatment of AIDS-related Kaposi's sarcoma and solid tumors (meeting abstract). Gill PS. Blood 1994;84(10, Suppl 1):248a